CLINICAL TRIAL: NCT03756701
Title: Mind Body Interventions for the Student Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Responsible Party: Principal Investigator, Nancy Landgraff, Professor, Youngstown State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 157-18
Record Dates: First submitted 2018-11-15; First posted 2018-11-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain; Anxiety; Stress
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: There will be 2 groups of participants. Group 1 will begin the intervention immediately. Group 2 will maintain their usual lifestyle for the first 10 weeks, and begin group sessions when group 1 has completed. There will be "refresher sessions" for group 1 once per month, and 3, 6 12 month follow up testing after the group sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Initial participants in the 10 mind body sessions
  Interventions: Behavioral: Mind body skills
- Group 2 (Active Comparator): 10 week no intervention groups - receives the mind body interventions after group 1 has completed.
  Interventions: Behavioral: Mind body skills

INTERVENTIONS:
Behavioral: Mind body skills — 2 hour skill sessions that focus on mindfulness: The topics for each session is based upon the Centers for Mind Body Medicine model. Both groups will follow this same weekly topic schedule.
  1. Introduction and Drawings
  2. Autogenic Training and Biofeedback
  3. Guided Imagery
  4. Meditation
  5. Mobilizing, Transforming, and Celebrating Emotion
  6. Genograms part 1
  7. Genograms part 2
  8. Mindful Eating and Healthy Nutrition
  9. Spirituality
  10. Closing Drawings and Ritual

SUMMARY:
This crossover randomized design study's objective is to see if mind body interventions can help students on a college campus manage their chronic pain and/or PTSD. Participants will attend 10 mind body skills group sessions that are 2 hours each. These group sessions teach a variety of ways (skills) for people to express their feelings. A licensed doctor, who is certified to teach mind-body skills group classes, will lead the skills group. Participants will be assessed with an anxiety questionnaire, a chronic pain measure and a measure of heart rate variability.

There will be two groups. Group 1 will begin intervention after baseline testing and will receive follow-up skill sessions once every month for 6 months. The first group will also attend bonus classes during the next 6 months. The second group will do baseline testing and no intervention for the first 10 weeks. They will then participate in the skills groups the second 10 weeks. There will be 3,6 and 12 month follow up data also taken.

DETAILED DESCRIPTION:
Students on campus will be made aware of the study through fliers posted on campus. If they contact the study representatives to participate, they will fill out a screening questionnaire that will determine their symptoms and care they are currently receiving. Those that meet the inclusion criteria will be assigned to Group 1 or 2 randomly. The mind body skills groups will be 10 weeks long. Group 1 will participate in mind body interventions immediately, and Group 2 will continue with their usual care for the 10 weeks. After the first session, Group 2 will complete the mind body intervention sessions. The research will therefore be a crossover randomized design where each group will serve as its own control, and also may be compared to the other group. Participants in either group will still be allowed to participate in any care they are currently receiving outside of the mind body intervention, including but not limited to counseling or a support group or therapy. Also, after these groups are over, the first group will continue to have "reunion groups" once per month for 6 months and the second group will not. Reunion groups will consist of supplementary mind body skills group sessions that reinforce skills learned in the original mind body skills groups and also work on retention of knowledge beyond the program. Outcome measures will be taken pre and post mind body skills group, and then at 3, 6, and 12 months after the 10 week mind body skills group ends.

The topics for each session is based upon the Centers for Mind Body Medicine model. Both groups will follow this same weekly topic schedule.

1. Introduction and Drawings
2. Autogenic Training and Biofeedback
3. Guided Imagery
4. Meditation
5. Mobilizing, Transforming, and Celebrating Emotion
6. Genograms part 1
7. Genograms part 2
8. Mindful Eating and Healthy Nutrition
9. Spirituality
10. Closing Drawings and Ritual

ELIGIBILITY:
Inclusion Criteria: Selection criteria includes:

Students aged 18-65 who own a smartphone that is able to download the HRV4Training app.

Students must be enrolled in graduate or undergraduate classes on Youngstown State University's campus.

Exclusion Criteria: students that have had previous experience with mind body skills groups or stress reduction interventions within the past 12 months.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Post Traumatic Stress Disorder Checklist - Civilian (PCLC) | Pre intervention, post intervention, 3,6,12 month followup
  Questionnaire
Change in Graded Chronic Pain Scale | Pre intervention, post intervention, 3,6,12 month followup
  Questionnaire
Change in Patient Health Questionnaire - 9 (PHQ 9), | Pre intervention, post intervention, 3,6,12 month followup
  Questionnaire
Change in Five Facet Mindfulness Questionnaire - 15 (FFMQ - 15) | Pre intervention, post intervention, 3,6,12 month followup
  Questionnaire
Change in Heart rate variability | Pre intervention, post intervention, at the start of each session, 3,6,12 month followup
  Measure of heart rate change over time taken with an ap on a cell phone.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Landgraff, PhD, Principal Investigator — Youngstown State University
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brennstuhl MJ, Tarquinio C, Montel S. Chronic Pain and PTSD: Evolving Views on Their Comorbidity. Perspect Psychiatr Care. 2015 Oct;51(4):295-304. doi: 10.1111/ppc.12093. Epub 2014 Nov 24. PMID 25420926
- [Background] Libby DJ, Pilver CE, Desai R. Complementary and Alternative Medicine Use Among Individuals with Posttraumatic Stress Disorder. Psychol Trauma. 2013;5: 277-285.
- [Background] Robert-McComb JJ, Cisneros A, Tacon A, Panike R, Norman R, Qian XP, McGlone J. The Effects of Mindfulness-Based Movement on Parameters of Stress. Int J Yoga Therap. 2015;25(1):79-88. doi: 10.17761/1531-2054-25.1.79. PMID 26667291
- See also: website — https://www.ptsd.va.gov/public/PTSD-overview/basics/how-common-is-ptsd.asp
- See also: website — https://www.psychiatry.org/patients-families/ptsd/what-is-ptsd